CLINICAL TRIAL: NCT06827769
Title: Study of Serum Zinc and Magnesium as Trace Elements in Patients With Chronic Liver Disease
Brief Title: Serum Zinc and Serum Magnesium in Chronic Liver Disease Patients
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Rania Mamdouh Elkafoury, Lecturer of Tropical medicine, Tanta University
Other Study IDs: 36264PR580/2/24
Record Dates: First submitted 2025-02-04; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Chronic Liver Disease and Cirrhosis
Keywords: serum zinc,; serum magnesium; chronic liver disease; cirhosis; trace elements
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: 60 healthy subjects as control.
  Interventions: Diagnostic Test: serum zinc and magnesium
- Chronic liver disease: 80 patients with chronic liver disease diagnosed by physical examination, laboratory investigations, and imaging study.
  This group will be subdivided into non-cirrhotic and cirrhotic liver groups.
  Interventions: Diagnostic Test: serum zinc and magnesium

INTERVENTIONS:
Diagnostic Test: serum zinc and magnesium — participants will be subjected to laboratory investigations (complete blood picture, liver and kidney function tests, Prothrombin time, international normalized ratio (INR), serum zinc, and magnesium).

SUMMARY:
The goal of this observational cross-sectional study is to assess the relationship between serum levels of magnesium and zinc in pediatric and adult patients with chronic liver disease and the clinic-laboratory variables.

Researchers will compare serum levels of zinc and magnesium in patients with chronic liver disease and healthy controls. Assess the correlation between serum zinc and magnesium and the presence and severity of chronic liver disease and cirrhosis.

Participants will be subjected to history taking, clinical examination, laboratory investigations, and abdominal ultrasonography.

DETAILED DESCRIPTION:
The progressive deterioration of liver tissue over time is a hallmark of chronic liver disorders (CLD). Liver diseases are linked to a number of risk factors, including environmental pollutants, genetics, and infectious diseases. The process of liver damage may be accelerated when multiple factors work together.

Due to their involvement in numerous metabolic pathways, trace elements are essential for preserving health. The liver plays a crucial role in controlling the metabolic pathway and transport, tissue distribution, toxicity, and trace element bioavailability. Certain metabolic illnesses are brought on by an excess or a shortage of certain trace elements, such as copper (Cu), magnesium (Mg), and zinc (Zn).

Zinc is necessary for DNA synthesis, RNA transcription, cell growth, protein synthesis, and regeneration. It also serves as a center of activity or cofactor for hundreds of enzymes (5). Numerous symptoms, such as anemia, dermatitis, stomatitis, alopecia, bedsores, decreased appetite, stunted growth, gonadal dysfunction, infection susceptibility, and taste problems, are brought on by zinc deficiency. Reduced albumin synthesis, low oral intake, increased urine excretion of zinc linked to portosystemic shunt, and impaired intestinal absorption are the causes of zinc insufficiency in CLD patients.

Magnesium is the fourth most abundant cation and the most prevalent intracellular ion. It has been connected to more than 300 enzymatic processes, including the cytolysis of antibodies, the synthesis of immunoglobin, and the adherence of resistant cells. Conversely, low magnesium levels in serum and liver tissue can slow the development of these conditions by interfering with mitochondrial activity, triggering inflammatory reactions, or causing metabolic anomalies.

This study aims to measure serum levels of zinc and magnesium in patients with chronic liver disease and to evaluate their correlation with clinic-laboratory variables.

This observational cross-sectional study will be performed on 80 subjects from the outpatient clinic and inpatient of the Tropical Medicine and Infectious Diseases Department and Pediatric Department at Tanta University Hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Chronic liver disease diagnosed by physical examination, laboratory investigations, and imaging study.

Exclusion Criteria:

1. Patients with Wilson disease.
2. Patients with chronic renal diseases.
3. Patients with IBD or any other cause of chronic diarrhea.
4. Drugs affecting levels of trace elements e.g. corticosteroids, digoxin thiazide, diuretics, and supplements 30 days before study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: subjects from the outpatient clinic and inpatient of the Tropical Medicine and Infectious Diseases Department and Pediatric Department at Tanta University Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
measuring serum zinc level in chronic liver disease patients | through study completion, an average of 1 year
measuring serum magnesium level in chronic liver disease patients | through study completion, an average of 1 year

SECONDARY OUTCOMES:
correlation of serum zinc and magnesium with liver disease severity | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Eman B Elsaadany, Principal Investigator — Pediatric medicine Department, Faculty of Medicine, Tanta University
Locations (1):
- Tanta University Hospitals, Tanta, Gharbyea, Egypt

IPD SHARING:
Plan to Share IPD: No